CLINICAL TRIAL: NCT07398352
Title: Comparison Of The Effect Of Interscalene Block Alone And The Combination Of Interscalene Block And Superficial Cervical Block On Brain Oxygenation And Carotid Artery Diameter In Shoulder Surgery
Brief Title: Comparison Of The Effects Of Regional Anesthesia On Brain And Carotid Artery Oxygenation In Shoulder Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, RAMAZAN ASLANPARÇASI, Specialist Of Anesthesiology And Reanimation, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISBSPBBO25
Record Dates: First submitted 2025-12-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Interscalene Block; Superficial Cervical Block; Cerebral Perfusion; Shoulder Surgeries
Keywords: brain perfusion; carotid artery diameter; interscalene brachial plexus block; superficial cervical plexus block; shoulder surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interscalene brachial plexus block (Active Comparator): The effect of interscalene block on cerebral perfusion and carotid diameter in shoulder surgery
  Interventions: Procedure: Interscalene brachial plexus block
- Combination of superficial cervical plexus block and interscalene brachial plexus block. (Experimental): Effects of combined interscalene block and superficial cervical block on cerebral perfusion and carotid diameter in shoulder surgery
  Interventions: Procedure: Interscalene brachial plexus block and superficial cervical plexus block

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — After sedating the patient with 2 mg midazolam, baseline values will be obtained, and an interscalene block will be performed under ultrasound guidance.
  Before the block, rSO2 values of both hemispheres of the brain and carotid artery diameter (at T1 and T5 times) will be measured and recorded using a NIRS probe at T2: 5 minute(min), T3: 10 min, T4: 15 min, and T5: 20 min.
  To assess the quality of the block, the sensory block will be evaluated at 20 minutes. The patient will be placed in a supine position, and after the first rSO2 value is obtained at T6, rSO2 values will be recorded at T7: 10 min, T8: 30 min, T9: 60 min, T10: surgical completion, and T11: 5 min postoperatively in the supine position. Bilateral carotid diameter(mm) will be measured at T6, T10, and T11. Before any postoperative analgesia is administered, the time of the patient's first pain and their need for analgesic will be recorded.
  Arms: interscalene brachial plexus block
Procedure: Interscalene brachial plexus block and superficial cervical plexus block — After sedating the patient with 2 mg midazolam, baseline values will be obtained, and a combined interscalene and superficial cervical block will be performed under ultrasound guidance.
  Before the block, rSO2 values of both hemispheres of the brain and carotid artery diameter(mm) (at T1 and T5 times) will be measured and recorded using a NIRS probe at T2: 5 minute, T3: 10 minute, T4: 15 minute, and T5: 20 minute.
  To assess the quality of the block, the sensory block will be evaluated at 20 minutes. The patient will be placed in a supine position, and after the first rSO2 value is obtained at T6, rSO2 values will be recorded at T7: 10 minute, T8: 30 minute, T9: 60 minute, T10: surgical completion, and T11: 5 minute postoperatively in the supine position. Bilateral carotid diameter(mm) will be measured at T6, T10, and T11. Before any postoperative analgesia is administered, the time of the patient's first pain, and their need for analgesic will be recorded.
  Other Names: interscalene block and superficial cervical plexus block
  Arms: Combination of superficial cervical plexus block and interscalene brachial plexus block.

SUMMARY:
The aim of our study was to compare the effects of interscalene block alone and the combination of interscalene block and superficial cervical block on cerebral oxygenation, carotid artery diameter, intraoperative hemodynamics, laboratory parameters, clinical course and postoperative pain in patients undergoing shoulder surgery.

DETAILED DESCRIPTION:
This study aimed to compare the effects of interscalene block alone and interscalene block combined with superficial cervical plexus block on cerebral oxygenation, carotid artery diameter, intraoperative hemodynamics, and postoperative pain in patients undergoing shoulder surgery.

Peripheral nerve blocks, particularly interscalene block, are commonly used in shoulder surgery due to their superior analgesic efficacy. Cerebral oxygenation was assessed using near-infrared spectroscopy (NIRS), a non-invasive method that reflects regional tissue oxygenation. The effects of both block techniques on bilateral cerebral oxygenation and carotid artery diameter were evaluated using NIRS and ultrasonography, respectively

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years patient
* American Society of Anesthesiologists (ASA) I-II patient

Exclusion Criteria:

* Age < 18 years or > 65 years
* History of carotid endarterectomy
* History of cerebrovascular accident(CVA)
* Body Mass index (BMI)>35 kg/m²
* Inability to cooperate or comply with study procedures
* Liver and kidney failure
* Pregnancy and breastfeeding
* ASA pyhsical status III-V
* Contraindication to regional anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The effect of regional anesthesia on cerebral oxygenation | Before block; T1 After block; T2: 5. minute, T3: 10. minute, T4: 15 minute, T5: 20 minute / In the beach chair position; T6: 1. minute, T7: 10. minute, T8: 30. minute, T9: 60. minute, T10: surgical end, Postoperative supine; T11: 5. minute
  We plan to investigate the effect of interscalene block or a combination of interscalene and superficial cervical block on oxygenation of both hemispheres of the brain using a NIRS probe.

SECONDARY OUTCOMES:
The effect of regional anesthesia on carotid artery diameter | Before block; T1 After block; T2: 5. minute, T3: 10. minute, T4: 15 minute, T5: 20 minute / In the beach chair position; T6: 1. minute, T7: 10. minute, T8: 30. minute, T9: 60. minute, T10: surgical end, Postoperative supine; T11: 5. minute
  The diameter of the common carotid artery will be measured longitudinally in millimeters(mm) with the transverse probe of the ultrasound at specified times.
The effect of the two-block method on the duration of first postoperative analgesia requirement and opioid consumption | From the end of surgery until the first request for postoperative analgesia and the amount of opioid comsumption, assessed up to 24 hours postoperatively
  The patient will not receive routine analgesia postoperatively. The time(hour) of the first request for analgesia and the amount of opioid consumption within the first 24 postoperative hours will be evaluated.

OTHER OUTCOMES:
Effect of block type on saturation | Before block; T1 After block; T2: 5. minute, T3: 10. minute, T4: 15 minute, T5: 20 minute / In the beach chair position; T6: 1. minute, T7: 10. minute, T8: 30. minute, T9: 60. minute, T10: surgical end, Postoperative supine; T11: 5. minute
  Peripheral oxygen saturation will be measured noninvasively from the finger using pulse oximetry.
Effect of block type on blood pressure | Before block; T1 After block; T2: 5. minute, T3: 10. minute, T4: 15 minute, T5: 20 minute / In the beach chair position; T6: 1. minute, T7: 10. minute, T8: 30. minute, T9: 60. minute, T10: surgical end, Postoperative supine; T11: 5. minute
  Blood pressure will be measured noninvasively from the arm
Effect of block type on heart rate | Before block; T1 After block; T2: 5. minute, T3: 10. minute, T4: 15 minute, T5: 20 minute / In the beach chair position; T6: 1. minute, T7: 10. minute, T8: 30. minute, T9: 60. minute, T10: surgical end, Postoperative supine; T11: 5. minute
  Heart rate will be measured continuously using electrocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan ASLANPARÇASI, MD, Principal Investigator — Sanliurfa Mehmet Akif Inan Education and Research Hospital

IPD SHARING:
Plan to Share IPD: No
Ethics committee approval covers only aggregate data analysis; there is no permission to share individual participant data.

REFERENCES:
- [Background] Ahmadzadeh S, Naccari BP, Amedio LS, Koruna AE, Bass D, Shekoohi S, Kaye AD. Efficacy of Suprascapular Versus Interscalene Block for Post-Operative Pain Management in Shoulder Surgeries: A Narrative Review. Curr Pain Headache Rep. 2025 Dec 29;30(1):13. doi: 10.1007/s11916-025-01443-7. PMID 41457137
- [Background] Cosarcan SK, Gurkan Y, Dogan AT, Koyuncu O, Ercelen O. Could Interscalene Block Possibly be Protective Against Cerebral Ischemia During Shoulder Surgery in a Beach Chair Position? Cureus. 2021 Jul 31;13(7):e16773. doi: 10.7759/cureus.16773. eCollection 2021 Jul. PMID 34476141
- [Background] Kaye AD, Upshaw WC, Holley C, Bailey PD, Tassin JP, Frolov MV, Sudini S, Miller BC, Palowsky ZR, Kataria S, Ahmadzadeh S, Shekoohi S, Robinson CL. Overview and Comparison of Interscalene Block Techniques for Brachial Plexus Pain Management. Curr Pain Headache Rep. 2024 Dec 30;29(1):1. doi: 10.1007/s11916-024-01346-z. PMID 39739068